CLINICAL TRIAL: NCT00824681
Title: Sound Of Family Together (S.O.F.T.) Music Program: A Randomized-Controlled Study to Investigate the Effect of Music Therapy on the Coping and Adjustment of Children of Adults With Major Burns
Brief Title: Effect of Music Therapy on Families of Burn Patients
Acronym: MTS3
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Music therapist left position.
Sponsor: MetroHealth Medical Center (Other)
Collaborators: The Cleveland Music School Settlement (Other); Kulas Foundation (Other)
Responsible Party: Xueli Tan, The Cleveland Music School Settlement
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 06-00891
Record Dates: First submitted 2009-01-15; First posted 2009-01-19 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Burns
Keywords: Psychological adjustment of family; family of patients; children of patients; intensive care unit; burn; music therapy; music; music program; anxiety; coping; adjustment; psychological stressor; emotional stressor
MeSH Terms: conditions — Burns; Anxiety Disorders; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Sound Of Family Together (S.O.F.T.) Music Program
  Interventions: Behavioral: Sound Of Family Together (S.O.F.T.) Music Program
- 2 (Active Comparator): Non-Therapy Related Activities (NTRA)
  Interventions: Other: Non-Therapy Related Activities (NTRA)

INTERVENTIONS:
Behavioral: Sound Of Family Together (S.O.F.T.) Music Program — Audio compact disk containing songs, music, special messages, poems from children of adults with major burns
  Arms: 1
Other: Non-Therapy Related Activities (NTRA) — NTRA includes non-directed activities e.g. reading books/magazines, watching TV/movie in family lounge off the BICU, playing with toys, listening to music CDs/radio.
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the efficacy of music therapy in assisting with the coping and adjustment of children of adults with major burns. The investigators hypothesized that there will be a significant decrease in anxiety levels between those children who participated in music therapy compared to non-participants.

DETAILED DESCRIPTION:
The Sound Of Family Together (S.O.F.T.) Music Program was introduced on a 14-bed burn intensive care unit to provide an avenue for communication between adults with major burns and their children. In adherence with unit policies, children under the age of 16 are only allowed onto the unit under very special circumstances, e.g. patient is under DNR status. This restriction may translate into a prolong absence between the patients and their young children; which may result in emotional and psychological stress factors such as separation anxiety, feelings of abandonment, and rejection of the parent when the patient is being discharged to home. Children who participate in the S.O.F.T. Music Program will record and produce an audio CD for their hospitalized parent/grandparent. The contents of the CD might include original songs, poems, and special messages created by the children. Pre and post tests results will determine the efficacy of the program to decrease anxiety levels in the children.

ELIGIBILITY:
Inclusion Criteria:

* Child's age between 6 - 14 years
* Child or grandchild of patient
* Child with limited visitation
* Adequate hearing, with correction
* Consenting non-hospitalized adult family member (NHAFM) speak/read English
* Child speak/read English
* Major physical or mental illness or disability does not interfere with ability to communicate for both consenting NHAFM and child

Exclusion Criteria:

* Child's age below 6 years and above 14 years
* Not the child or grandchild of patient
* Child with unlimited visitation
* Hearing loss that interferes with ability to communicate
* NHAFM does not speak/read English
* Child does not speak/read English
* Major physical or mental illness or disability interferes with ability to communicate for both consenting NHAFM and child
* Patient on observation status, i.e. only one overnight stay

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Anxiety level | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xueli Tan, MM, MT-BC, Study Chair — The Cleveland Music School Settlement; Charles J Yowler, MD, FACS, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States